CLINICAL TRIAL: NCT03912480
Title: Study on the Efficacy and Safety of Stem Cells From Human Exfoliated Teeth in Treating Diabetic Patients With Significantly Reduced Islet Function
Brief Title: Stem Cells From Human Exfoliated Teeth in Treatment of Diabetic Patients With Significantly Reduced Islet Function
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CAR-T (Shanghai) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTLC002
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stem cells from human exfoliated teeth (Experimental): Basic treatment:
  The original treatment regimen was maintained. During the study period, insulin dose could be adjusted with the change of blood glucose, while the type and dose of oral hypoglycemic drugs remained unchanged (except when side effects of drugs or insulin preparations were stopped or patients still had frequent hypoglycemia).
  Stem cell therapy:
  Dosage: Stem cells from human exfoliated teeth were calculated at 0.11IU/kg body weight .
  Course of treatment: 3 times, Injections were administered at enrollment, 2 weeks after enrollment, and 6 weeks after enrollment.
  Note: at 1 month follow-up (V5) after the last transplantation of several cells, the subjects were still unable to discontinue insulin, and then began the second course of stem cell therapy.After the second course of treatment, the follow-up plan was resumed.
  Interventions: Biological: Stem cells from human exfoliated teeth

INTERVENTIONS:
Biological: Stem cells from human exfoliated teeth — Intravenous infusion of pulp mesenchymal stem cells

SUMMARY:
To evaluate the safety and efficacy of Stem cells from human exfoliated teeth transplantation in patients with Islet function decreased significantly to provides scientific basis for further clinical studies to verify the safety and efficacy. On the basis of maintaining the original treatment, intravenous drip of dental pulp mesenchymal stem cells.

DETAILED DESCRIPTION:
Basic treatment:

The original treatment regimen was maintained. During the study period, insulin dose could be adjusted with the change of blood glucose, while the type and dose of oral hypoglycemic drugs remained unchanged (except when side effects of drugs or insulin preparations were stopped or patients still had frequent hypoglycemia).

Stem cell therapy:

Dosage: Stem cells from human exfoliated teeth were calculated at 0.11IU/kg body weight .

Course of treatment: 3 times, Injections were administered at enrollment, 2 weeks after enrollment, and 6 weeks after enrollment.

Note: at 1 month follow-up (V5) after the last transplantation of several cells, the subjects were still unable to discontinue insulin, and then began the second course of stem cell therapy.After the second course of treatment, the follow-up plan was resumed.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the purpose of clinical trials, willing to participate and sign informed consent;
2. Patients with type 2 diabetes are clearly diagnosed according to WHO diagnostic criteria and whose disease duration is more than 5 years, or whose disease duration of type 1 diabetes is more than 1 year;
3. Islet function test (steamed bread test) : c-peptide fasting 1ng/ml, 2 hours 2ng/ml
4. Insulin (with or without oral hypoglycemic therapy) and fasting blood glucose (FPG)9.0mmol/L, HbAlc 8.5; The service life of oral hypoglycemic drugs (including metformin, alpha-glucosidase inhibitors or insulin secreting agents) was more than 3 months.
5. Age 25-70 years old, gender not limited;
6. Body mass index (BMI) : between 19 and 28kg/m2;
7. from the date of screening to the end of follow-up, male or female subjects of childbearing age will voluntarily take precautions Pregnancy; Urine pregnancy test was negative when screening women of childbearing age, and serum pregnancy test was performed when necessary to clearly exclude pregnancy.-

Exclusion Criteria:

1. Patients with gestational diabetes or other special types of diabetes;
2. Acute complications such as diabetic ketoacidosis and non-ketotic hyperosmolar syndrome were screened within the first month;
3. Patients who have received other stem cell therapy before screening;
4. Blood pressure of patients with poor blood pressure control: 160/100mmhg at the time of screening;
5. Those who took thiazolidinediones, ddp-iv inhibitors and glp-1 drugs within the first 3 months were screened;
6. Patients who have used insulin for less than 1 year before screening and only injected insulin subcutaneously once a day within the past 3 months;
7. Patients with pancreatic diseases, including those with acute and chronic pancreatitis and pancreatic tumors;
8. Patients with other malignant tumors or suspected tumor tendency;Or in the active phase of various infections (including active stage of HBV or HCV infection);Immunodeficiency virus (HIV) positive patients;
9. Patients with other serious systemic diseases (such as cardiovascular system, respiratory system, digestive system, nervous system, endocrine system, urogenital system, immune system and blood system);
10. For patients with liver and kidney dysfunction, for example, serum bilirubin TBIL exceeds 1.5 times of the normal upper limit, AST and ALT exceed 2.5 times of the normal upper limit, and serum creatinine Cr exceeds 1.2 times of the normal upper limit;
11. Is on systemic sex hormone (glucocorticoid), immunosuppressant or cytotoxic therapy;
12. Disabled patients (blind, deaf, dumb, mentally retarded, physically disabled) as stipulated by law, pregnant women and lactating women;People suffering from mental illness;Patients who take drugs or have a history of adverse drug abuse and alcohol dependence within 5 years;
13. Patients with contraindications or allergies treated in this study;
14. Subjects who have participated in other clinical studies in the past 3 months.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-01-05 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Total daily insulin dose | baseline and 1,2,6 week and 2,3,6,9,12 month
  change from baseline during treatment
glucose-c peptide release test | baseline and 1,2,6 week and 2,3,6,9,12 month
  relative baseline change during treatment

SECONDARY OUTCOMES:
Islet function | 1 year
  c-peptide and proinsulin
Composite index of glycosylated hemoglobin (HbAlc) and frequency of hypoglycemia | 1 year
  Changes relative to baseline during treatment
Continuous dynamic blood glucose | 1 year
  Changes relative to baseline during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Qin Huang, Doctor, Principal Investigator — Changhai houspital
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China